CLINICAL TRIAL: NCT07068802
Title: Message Framing in HPV Vaccination Decision: A Survey Experimental Study Among Chinese Male College Students
Brief Title: Message Framing in HPV Vaccination Decision
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zhejiang University (Other)
Responsible Party: Principal Investigator, Bo Yan, professor, Zhejiang University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 20240010
Record Dates: First submitted 2025-07-07; First posted 2025-07-16 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: HPV Vaccination Intention Among Male College Students
Keywords: HPV; VACCINE; COMMUNICATION; INTENTION
MeSH Terms: conditions — Communication

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: The study is double-blinded, meaning that both the subjects and the researchers are unaware of the group assignments. The randomization of groups is conducted using Wenjuanxing (a survey tool). However, blinding is not implemented during data analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- control group (Active Comparator): HPV risks
  Interventions: Behavioral: Message framing
- intervention group 1 (Experimental): HPV risks+personal risks
  Interventions: Behavioral: Message framing
- intervention group 2 (Experimental): HPV risks+partner risks
  Interventions: Behavioral: Message framing
- intervention group 3 (Experimental): HPV risks+personal risks and partner risks
  Interventions: Behavioral: Message framing

INTERVENTIONS:
Behavioral: Message framing — Participants provided electronic informed consent with voluntary withdraw options. Randomization was implemented through a 1:1:1:1 allocation ratio to four conditions: Control group (Group 1, n=154) receiving a standard statement of HPV risks (In mainland China, HPV vaccines are currently approved only for female use. However, in other countries, they are also available for males. HPV can cause cancers throughout the body, from the head to the reproductive system. Thus, HPV vaccination can protect against many cancer types. Annually, over 120,000 Chinese are diagnosed with HPV-related cancers, with about 50,000 dying from them.); Intervention 1 (Group 2, n=152) adding male-specific health risks; Intervention 2 (Group 3, n=153) adding risk to female partners; Intervention 3 (Group 4, n=153) adding both personal risk and risk to female partners. The protocol involved sequential completion of pre-exposure questionnaires, timed 120-second message exposure, and immediate post-exposure asses

SUMMARY:
The goal of this clinical trial is to determine if different risk communication strategies can increase the intention to receive the HPV vaccine among male college students in China. The study focuses on male college students aged 18-25 years, who are healthy volunteers and have not previously received the HPV vaccine. The main question it aims to answer is:

Can specific risk communication interventions increase the willingness to receive the HPV vaccine among male college students?

Researchers will compare four different interventions to see if they have a significant effect on vaccination intention:

Control group: Receiving a standard statement about HPV risks. Personal risks group: Receiving information on male-specific health risks. Partner risks group: Receiving information on risks to female partners. Combined risks group: Receiving information on both personal risks and risks to female partners.

Participants will:

Provide electronic informed consent. Complete pre-exposure questionnaires. Be exposed to a 120-second message based on their assigned group. Complete an immediate post-exposure assessment. This study aims to identify effective communication strategies to promote HPV vaccination among male college students, especially in light of the upcoming approval of the first male HPV vaccine in China.

DETAILED DESCRIPTION:
Study design We conducted a randomized survey experiment with pre-post design between December 2024 to January 6th 2025, right before the approval of the first HPV vaccine for male in the country in January 8th across three geographically dispersed Chinese universities (eastern, western, and northern regions). This study was conducted from The Institutional Review Board of Hangzhou Normal University, School of Public Health approved this study (approval no. 20240010).

Participants The proportion of male college students intending to receive the HPV vaccine was assumed to be 45% in the calculation of sample size, based on a previous report in China [28]. We assumed an increase in vaccination willingness to 55% for the personal risks group and partner risks group and 65% for the both risks group. To detect a significant intervention effect with a 2-sided α = .05, a power of 0.80, and an 80% valid response rate, we calculated that 169 participants were required (676 participants total).

From 720 initially involved in baseline evaluation, we excluded 82 due to incompleteness (>10% missing data) or invalidity (i.e., inconsistent responses to attention-check items), and 35 additional participants reporting prior HPV vaccination or definite baseline vaccination intention, yielding a final analytical sample of 612 male college students.

Randomization and interventions Participants provided electronic informed consent with voluntary withdraw options. Randomization was implemented through a 1:1:1:1 allocation ratio to four conditions: Control group (Group 1, n=154) receiving a standard statement of HPV risks (In mainland China, HPV vaccines are currently approved only for female use. However, in other countries, they are also available for males. HPV can cause cancers throughout the body, from the head to the reproductive system. Thus, HPV vaccination can protect against many cancer types. Annually, over 120,000 Chinese are diagnosed with HPV-related cancers, with about 50,000 dying from them.); Intervention 1 (Group 2, n=152) adding male-specific health risks; Intervention 2 (Group 3, n=153) adding risk to female partners; Intervention 3 (Group 4, n=153) adding both personal risk and risk to female partners. The protocol involved sequential completion of pre-exposure questionnaires, timed 120-second message exposure, and immediate post-exposure assessment.

Measures We evaluated three primary outcomes. The first outcome is vaccination intention ("If HPV vaccine were available for males in China, would you get vaccinate?"). The answer was measured using a 5-point Likert scale (1= "not at all willing" to 5= "highly willing") and then dichotomized into "willing (4-5)" vs. "unwilling (1-3)". The second outcome is Precaution Adoption Process Model (PAPM) adapted decisional readiness. A single question was asked "Before today, what do your stance on HPV vaccination?" the answer was categories as "pre-decisional (never heard/knew but no consideration) vs. "decisional (active refusal/acceptance). The third outcome aims to test the respondents' perceived responsibility toward HPV infection prevention with a single question "HPV infection is a shared responsibility of both genders." The answer was measured using a 5-point Likert scale on agreement (1= "strongly disagree" to 5= "strongly agree"). The final answer was dichotomized into "agree (4-5)" and "disagree (1-3)".

Statistical analysis Chi-square test and Kruskal-Wallis H test were performed to compare the frequencies and percentages of participants' demographic characteristics across groups. McNemar's test and Chi-square test were used to compare the effect within and between groups respectively. Multivariate logistic regression models, adjusting for sociodemographic factors (e.g., age and education background), were adopted to evaluate the differences between the four groups. All statistical analyses were performed using SPSS version 27.0, based on different statistical significance levels of p value after Bonferroni correction.

ELIGIBILITY:
Inclusion Criteria:

- aged above 18, male,college student, willing to participate

Exclusion Criteria:

- vaccinated with one dose or more HPV vaccine or decided to get vaccinated with HPV vaccine.

Ages: 18 Years to 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 612 (Actual)
Dates: Start 2024-12-10 (Actual); Primary Completion 2025-01-06 (Actual); Study Completion 2025-01-06 (Actual)

PRIMARY OUTCOMES:
HPV vaccination intention | Immediately after the 120-second message exposure.
  The primary outcome measure is the intention to receive the HPV vaccine among male college students, assessed through a question: "If HPV vaccine were available for males in China, would you get vaccinate?". The answer was measured using a 5-point Likert scale (1= "not at all willing" to 5= "highly willing")
Precaution Adoption Process Model (PAPM) adapted decisional readiness | Immediately after the 120-second message exposure.
  A single question was asked "Before today, what do your stance on HPV vaccination?" the answer was categories as "pre-decisional (never heard/knew but no consideration) vs. "decisional (active refusal/acceptance).
respondents' perceived responsibility toward HPV infection prevention | Immediately after the 120-second message exposure.
  The third outcome aims to test the respondents' perceived responsibility toward HPV infection prevention with a single question "HPV infection is a shared responsibility of both genders." The answer was measured using a 5-point Likert scale on agreement (1= "strongly disagree" to 5= "strongly agree").

CONTACTS AND LOCATIONS:
Locations (1):
- Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Yes